CLINICAL TRIAL: NCT05171751
Title: Beijing Children's Hospital, Capital Medical University, National Center for Children's Health
Brief Title: Efficacy and Safety Evaluation of Octreotide in the Treatment of Congenital Hyperinsulinemia
Acronym: BCH
Status: Completed | Type: Observational
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Chunxiu Gong, director, Beijing Children's Hospital
Other Study IDs: octreotide-CHI-2021
Record Dates: First submitted 2021-11-05; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Congenital Hyperinsulinaemic Hypoglycaemia; Octreotide Adverse Reaction
MeSH Terms: interventions — Octreotide; Glucose

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Octreotide Injection — Octreotide subcutaneous injection for congenital hyperinsulinemia with ineffective diazine
  Other Names: glucose

SUMMARY:
To analyze and evaluate the efficacy and safety of octreotide subcutaneous injection in the treatment of diazazine-ineffective congenital hyperinsulinemia (CHI) in children.

DETAILED DESCRIPTION:
Octreotide subcutaneous injection is effective and safe in the treatment of congenital hyperinsulinemia in children with inefficacy of diazazine.

ELIGIBILITY:
Inclusion Criteria:

1. Consistent with the diagnosis of congenital hyperinsulinemia with ineffective diazine; With the maximum dose of diazine at 15mg/kg/d for 5 days, fasting blood glucose/postprandial blood glucose could not be stabilized at the target value of 3.3mmol/L without intravenous glucose infusion.
2. patients treated with octreotide subcutaneous injection.

Exclusion Criteria:

1. Before the diagnosis of CHI and the treatment related to CHI, the child had received total pancreatectomy without octreotide
2. Secondary hypoglycemia caused by diseases other than CHI
3. Patients who refused to take octreotide due to parents or family economic reasons, but not hospital treatment factors.
4. Patients who intervene/interfere with octreotide treatment regimen for parental reasons

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with congenital hyperinsulinemia who received octreotide subcutaneous injection after diazazine treatment failed.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
blood glucose | 1 year
  Maintain target blood glucose ≥3.3mmo/L

CONTACTS AND LOCATIONS:
Overall Officials: bingyan cao, doctor, Principal Investigator — doctor of Beijing children's hospital
Locations (1):
- Department of Endocrinology, Genetics, Metabolism, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided